CLINICAL TRIAL: NCT05177120
Title: Central Sensitization in Familial Mediterranean Fever: A Cross-Sectional Observational Study
Brief Title: Central Sensitization in Familial Mediterranean Fever (FMF)
Acronym: FMF
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 06.12.2019.1053
Record Dates: First submitted 2022-01-03; First posted 2022-01-04 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2021-12

CONDITIONS: Familial Mediterranean Fever; Central Sensitisation
Keywords: Familial Mediterranean Fever; Central Sensitization; Central Sensitization Inventory
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — ametantrone; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FMF patients: Patients with diagnosed FMF
  Interventions: Diagnostic Test: Central Sensitization Inventory; Other: Short form-36; Other: Pittsburgh Sleep Quality Index; Other: Health assessment questionnaire; Other: Hospital anxiety and depression scale; Diagnostic Test: Fibromyalgia rapid screening tool; Other: Familial Mediterranean Fever Quality of life scale

INTERVENTIONS:
Diagnostic Test: Central Sensitization Inventory — Standardized questionnaire to determine the level of central sensitization
  Other Names: CSI
Other: Short form-36 — Standardized questionnaire to investigate the quality of life in patients
  Other Names: SF-36
Other: Pittsburgh Sleep Quality Index — Standardized questionnaire to investigate the sleep quality and disturbance
  Other Names: PSQI
Other: Health assessment questionnaire — Standardized questionnaire used to detect the presence of disability
  Other Names: HAQ
Other: Hospital anxiety and depression scale — Standardized questionnaire to investigate the depression and anxiety
  Other Names: HADS
Diagnostic Test: Fibromyalgia rapid screening tool — Standardized questionnaire to determine the presence of fibromyalgia
  Other Names: FIRST
Other: Familial Mediterranean Fever Quality of life scale — Standardized questionnaire to investigate the quality of life in Familial Mediterranean Fever patients
  Other Names: FMFQoL

SUMMARY:
Familial Mediterranean Fever (FMF) is an autosomal recessive inherited disease with a course of autoinflammation, which is characterized by the episodes of fever and serositis. Central sensitization (CS) is defined as increased response to normal or sub-threshold stimuli of central nervous system and its close relationship with many rheumatological diseases has been demonstrated in several studies. However, there are no data on the frequency of CS in FMF patients.

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) is a self-limiting autoinflammatory disease with well-defined genetic and clinical features. Recurrent episodes of fever and serositis accompanied by increased acute phase reactants and good response to colchicine are the core components of the disease. The frequency of this disease, which is common in Eastern Mediterranean countries, is variable according to regions, but it is reported as 1/1000. In the pathogenesis of the disease, the mutation of the MEFV (Mediterranean Fever) gene, which is located on the 16th chromosome and encodes the pyrin protein, is known as the basic mechanism.In rheumatic diseases, inflammatory mediators cause CS by first creating changes in the regulation of pain in peripheral neurons and then in spinal and supraspinal pathways. Stimulation of peripheral nerves by mediators released during inflammation results in neurogenic inflammation, which is among the peripheral sensitization (PS) mechanisms. PS is defined as the increased sensitivity of nociceptive neurons to normal or below-threshold stimuli and constitutes the first step in the development of CS.Similar to other autoimmune diseases, it is possible that the neuroinflammatory process triggers peripheral and central sensitization mechanisms in FMF patients and affects pain pathways.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study

Exclusion Criteria:

* Had another systemic inflammatory rheumatic diseases
* Using centrally acting pain medications (e.g., pregabalin, duloxetine, opioids) or glucocorticoids (>10 mg prednisone or its equivalent)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with FMF
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | 6 months
  25 somatic and psychosocial symptoms, which are frequently found in patients with central sensitization in part A, are questioned. In part B, the presence of diseases whose relationship with central sensitization is well defined is questioned in the patient without participating in scoring. Central sensitization is assumed in patients who score 40 or more over 100 points.

SECONDARY OUTCOMES:
Short form-36 (SF-36) | 6 months
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health.The scale consists of 36 questions questioning 8 sub-parameters regarding the health status of the person.These parameters are physical function, pain, limitation due to physical and emotional problems, emotional well-being, social function, fatigue and general health perception. High scores are associated with improved quality of life.
Familial Mediterranean Fever Quality of Life Scale (FMF-QoL) | 6 months
  FMF-QoL was developed to evaluate the quality of life in FMF patients. This scale consists of 20 questions in the form of a Likert scale and the total scoring is between 0-80. High scores indicate a decrease in quality of life.
Health Assessment Questionnaire (HAQ) | 6 months
  n the scale, difficulty in performing 20 specific tasks from 8 categories is questioned and the scoring is between 0-60. High scores are associated with increased disability.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  This scale consists of 14 questions in total, and anxiety symptoms are questioned in half of the questions and depression-related complaints in the other half. A subscore of 8 or higher for depression or anxiety is considered a clinical case.
Pittsburgh Sleep Quality Index (PSQI) | 6 months
  The questionnaire includes 21 questions covering 7 components that investigate the symptoms of sleep disturbances. Scores range from 0 to 21 and a score of >5 is considered as a sleep disorder.
Fibromyalgia Rapid Screening Tool (FIRST). | 6 months
  This scale consists of 6 questions investigating the most relevant clinical features of fibromyalgia. The questions are answered as yes/no and 5 or more out of 6 points in total are in favor of fibromyalgia.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Sanal- Toprak, Asst.Prof, Study Chair — Marmara University
Locations (1):
- Feyza Nur Yücel, Sinop, Turkey (Türkiye)

REFERENCES:
- [Background] Lee YC, Bingham CO 3rd, Edwards RR, Marder W, Phillips K, Bolster MB, Clauw DJ, Moreland LW, Lu B, Wohlfahrt A, Zhang Z, Neogi T. Association Between Pain Sensitization and Disease Activity in Patients With Rheumatoid Arthritis: A Cross-Sectional Study. Arthritis Care Res (Hoboken). 2018 Feb;70(2):197-204. doi: 10.1002/acr.23266. PMID 28437846
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Pinar R. Reliability and construct validity of the SF-36 in Turkish cancer patients. Qual Life Res. 2005 Feb;14(1):259-64. doi: 10.1007/s11136-004-2393-3. PMID 15789959
- [Background] Unal-Ulutatar C, Duruoz MT. Development and validation of a quality of life scale in Familial Mediterranean Fever (FMFQoL). Mod Rheumatol. 2021 May;31(3):710-717. doi: 10.1080/14397595.2020.1775946. Epub 2020 Jun 26. PMID 32475195
- [Background] Senerdem N, Gul A, Konice M, Aral O, Ocal L, Inanc M, Yuzbasioglu N. The use of two different Health Assessment Questionnaires in Turkish rheumatoid arthritis population and assessment of the associations with disability. Clin Rheumatol. 1999;18(1):33-7. doi: 10.1007/s100670050048. PMID 10088946
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Familial Mediterranean fever (FMF) in Turkey: results of a nationwide multicenter study. Medicine (Baltimore). 2005 Jan;84(1):1-11. doi: 10.1097/01.md.0000152370.84628.0c. PMID 15643295
- [Background] Ancient missense mutations in a new member of the RoRet gene family are likely to cause familial Mediterranean fever. The International FMF Consortium. Cell. 1997 Aug 22;90(4):797-807. doi: 10.1016/s0092-8674(00)80539-5. PMID 9288758
- [Background] Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. J Pain. 2009 Sep;10(9):895-926. doi: 10.1016/j.jpain.2009.06.012. PMID 19712899
- [Background] Silva RL, Lopes AH, Guimaraes RM, Cunha TM. CXCL1/CXCR2 signaling in pathological pain: Role in peripheral and central sensitization. Neurobiol Dis. 2017 Sep;105:109-116. doi: 10.1016/j.nbd.2017.06.001. Epub 2017 Jun 3. PMID 28587921